CLINICAL TRIAL: NCT05634044
Title: eNose Validation Study: Correlating Volatile Organic Compounds With Daily Fiber Intake
Brief Title: Validating eNose Measurement of Daily Fiber Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Robin Voigt, Principle Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22041203-IRB01
Record Dates: First submitted 2022-11-15; First posted 2022-12-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Dietary Fiber

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eNose device use (Experimental): Participants will place the e-Nose device in their bathroom to record VOCs from the ambient air after they have a bowel movement. In addition to this, all participants will complete 2 blood draws 3 stool collections, and questionnaires over the course of 4 visits during a 3 week period.
  Interventions: Device: eNose Device

INTERVENTIONS:
Device: eNose Device — Participants will place the e-Nose device in their bathroom to record VOCs from the ambient air after they have a bowel movement. In addition to this, all participants will complete 2 blood draws 3 stool collections and questionnaires over the course of 4 visits during a 3-week period.

SUMMARY:
Monitoring dietary intake and digestion is important for both medical monitoring and assessing the wellness of individuals. Fiber is an important nutrient that is not focused on enough, despite it being an essential nutrient for the bacteria and other micro-organisms that reside in our GI Tracts, known as the microbiome. Ingestion of fermentable soluble and insoluble dietary fiber has been shown to result in the production of short-chain fatty acids (SCFA) by the colonic microbiome. These SCFAs are volatile organic compounds (VOCs) and can be detected in the atmosphere of a bowel movement. We have developed an e-Nose device that once placed in the bathroom records volatile organic compounds (VOCs) from the ambient air. We have demonstrated in an "N of 1" study a strong correlation between the eNose output and grams of daily fiber intake.

The current study is being proposed to validate the e-Nose device on a larger population. This is a nonmedical device that is not regulated by the FDA. A total of 40 subjects are invited to participate in this 3-week study. Participants will be asked to complete questionnaires and provide stool and blood samples. The subjects will place the eNose device in their bathroom and record their daily food intake over a 3-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 21-65, with no chronic medical diseases (mild and controlled hypertension, and controlled hyperlipidemia are acceptable).
2. Willingness to eat 2 prebiotic bar per day for two weeks and collect stool samples three times, provide blood samples twice and complete questionnaires.

Exclusion Criteria:

1. Patients on a restricted diet (e.g., gluten-free diet, Paleo diet, vegetarian or vegan diet)
2. Allergy to almonds, flax seed, or coconuts
3. Chronic GI disorders (Inflammatory bowel disease, Irritable Bowel Syndrome on regular therapy taking fiber or MiraLAX is acceptable to be enrolled; celiac disease, colon cancer, intestinal resection,)
4. Chronic NSAID use (more than 3 days per week)
5. Antibiotic use in the last 12 weeks
6. BMI > 35 or < 18
7. Inability to sign an informed consent form
8. Non-English speaker

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Accuracy of this device to detect increased intake of fiber | 3 weeks
  Assessed by comparing percentage change in volatile organic compounds (measured in OHMS) against the daily fiber intake in grams

SECONDARY OUTCOMES:
Ability of eNose to detect increased production of SCFA- positive correlation between enose signals and each of three SCFA and total SCFA levels in stool | 3 weeks
  Assessed by comparing eNose signal recordings (measured in OHMS) and each of three SCFA and total SCFA levels in stool
Impact of fiber bar in microbiota composition | 3 weeks
  Assessed by 16s amplicon and function- SCFA levels
Tolerability of prebiotic bar | 3 weeks
  Assessed by GI PROMIS questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States